CLINICAL TRIAL: NCT06255743
Title: (Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-Double Strad DNA Antibodies) Correlate With Depression and Anxiety in Systemic Lupus Erythematosus Patients
Brief Title: (Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-ds DNA Antibodies) and Relation to Depression and Anxiety in SLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Maher Kamaly, assistant lecture at rhematology and rehabilitation department at sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-01-07MD
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Depression -Anxiety-Anti-Ribosomal P Protein Antibody - Anti-U1 Antibody - Anti-Nucleosome Antibody - Anti-Double Strad DNA Antibody
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case (Experimental): cases diagnosed systemic lupus erythematosus we measure degree of depression and anxiety and relation to (Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-ds DNA Antibodies)
  Interventions: Diagnostic Test: Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-Double Strad DNA Antibodies

INTERVENTIONS:
Diagnostic Test: Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-Double Strad DNA Antibodies — determine Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-Double Strad DNA Antibodies) and its relation to the degree of Depression and Anxiety in Systemic Lupus Erythematosus Patients

SUMMARY:
the study determine the relation between the degree of (Depression and Anxiety) in Systemic Lupus Erythematosus Patients by zung self rating depression scale and zung self rating anxiety scale and (Anti-Ribosomal P Protein,Anti-U1 RNP, Anti-Nucleosome and Anti-Double Strad DNA Antibodies).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfill the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria or 2019 American College of Rheumatology/European League against Rheumatism classification criteria of Systemic Lupus Erythematosus.
2. Patients who is able to give informed consent to join the study.

Exclusion Criteria:

* - Any patient with any autoimmune disease other than systemic lupus erythematosus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-14 (Estimated); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
the degree of depression | 1 year
  by using zung self-rating depression scale
the degree of anxiety | 1 year
  by using zung self-rating anxiety scale

SECONDARY OUTCOMES:
Anti-Ribosomal P Protein antibody | 1 year
  was examined by ANA profile by immunoblot based assay with which the plasma of heparin-anticoagulated venous blood and there of IgG antibodies reacted against the auto-antigens are tested.
Anti-U1 RNP antibody | 1 year
  was examined by ANA profile by immunoblot based assay with which the plasma of heparin-anticoagulated venous blood and there of IgG antibodies reacted against the auto-antigens are tested.
Anti-Nucleosome antibody | 1 year
  was examined by ANA profile by immunoblot based assay with which the plasma of heparin-anticoagulated venous blood and there of IgG antibodies reacted against the auto-antigens are tested.
Anti-Double Strad DNA Antibody | 1 year
  was examined by ANA profile by immunoblot based assay with which the plasma of heparin-anticoagulated venous blood and there of IgG antibodies reacted against the auto-antigens are tested.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amoura Z, Koutouzov S, Chabre H, Cacoub P, Amoura I, Musset L, Bach JF, Piette JC. Presence of antinucleosome autoantibodies in a restricted set of connective tissue diseases: antinucleosome antibodies of the IgG3 subclass are markers of renal pathogenicity in systemic lupus erythematosus. Arthritis Rheum. 2000 Jan;43(1):76-84. doi: 10.1002/1529-0131(200001)43:13.0.CO;2-I. PMID 10643702
- [Background] Benito-Garcia E, Schur PH, Lahita R; American College of Rheumatology Ad Hoc Committee on Immunologic Testing Guidelines. Guidelines for immunologic laboratory testing in the rheumatic diseases: anti-Sm and anti-RNP antibody tests. Arthritis Rheum. 2004 Dec 15;51(6):1030-44. doi: 10.1002/art.20836. No abstract available. PMID 15593352
- [Background] Diamond B, Bloom O, Al Abed Y, Kowal C, Huerta PT, Volpe BT. Moving towards a cure: blocking pathogenic antibodies in systemic lupus erythematosus. J Intern Med. 2011 Jan;269(1):36-44. doi: 10.1111/j.1365-2796.2010.02318.x. PMID 21158976
- [Background] Schattner E, Shahar G, Lerman S, Shakra MA. Depression in systemic lupus erythematosus: the key role of illness intrusiveness and concealment of symptoms. Psychiatry. 2010 Winter;73(4):329-40. doi: 10.1521/psyc.2010.73.4.329. PMID 21198385
- [Background] Gao HX, Campbell SR, Cui MH, Zong P, Hee-Hwang J, Gulinello M, Putterman C. Depression is an early disease manifestation in lupus-prone MRL/lpr mice. J Neuroimmunol. 2009 Feb 15;207(1-2):45-56. doi: 10.1016/j.jneuroim.2008.11.009. Epub 2009 Jan 3. PMID 19121871